CLINICAL TRIAL: NCT04456036
Title: Rehabilitation Needs and Functional Recovery in Covid-19 Acute and Post-acute Care: Study of Functional Evolution, Predictors of Activities and Participation Recovery After Severe Covid-19 and Rehabilitation Role
Brief Title: Rehabilitation Needs and Functional Recovery in Covid-19 Acute and Post-acute Care
Acronym: RECOVER-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Università Politecnica delle Marche (Other)
Collaborators: Maria Gabriella Ceravolo (Unknown); Michela Coccia (Unknown); Lauredana Ercolani (Unknown); Elisa Andrenelli (Unknown); Lucia Pepa (Unknown); Rossella Cima (Unknown); Michela Aringolo (Unknown)
Responsible Party: Principal Investigator, Marianna Capecci, PhD, Prof, Università Politecnica delle Marche
Other Study IDs: NeuroRehabAN_Covid_2020
Record Dates: First submitted 2020-06-30; First posted 2020-07-02 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: COVID-19
Keywords: COVID-19; Rehabilitation; Recovery of Function; Activities of Daily Living; Prognosis; Quality of Life; Continuity of Patient Care
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to apply a prospective observational design to describe the emerging functional impairments of subjects affected by COVID-19 in the acute phase and monitor their course and impact on activities and participation up to 12 months of onset. The ultimate goal is to provide a reliable framework to plan rehabilitation delivery to COVID-19 survivors in each phase and foresee health needs in the medium and long term. The secondary objective of the study is to find predictors of functional recovery, among pre-existing and emerging individual and contextual factors, with a special focus on the latency of rehabilitation start after hospital admission.

DETAILED DESCRIPTION:
The disease caused by SARS-CoV-2 infection, COronaVIrus Disease-19 (COVID-19), was first reported on December 31, 2019. About 20% patients, mostly elderly people, suffered from a severe form of acute respiratory failure. COVID-19 is a new clinical entity, therefore its understanding is largely incomplete, in particular as regards medium and long term consequences both in the clinical and functional domain. An early integration of rehabilitation care since the acute phase is often required to cope with the functional sequelae of the severe respiratory syndromes, as well of cardiac and neurological complications. However, indications, approaches, timing, amount and settings are mainly unknown due to the lack of epidemiological data regarding the impact of COVID-19 in terms of body function impairment and activity limitations in the short term and participation restrictions in the medium and long-term.

The purpose of the study is to apply a prospective observational design to describe the emerging functional impairments of subjects affected by COVID-19 in the acute phase and monitor their course and impact on activities and participation up to 12 months of onset. The ultimate goal is to provide a reliable framework to plan rehabilitation delivery to COVID-19 survivors in each phase and foresee health needs in the medium and long term. The secondary objective of the study is to find predictors of functional recovery, among pre-existing and emerging individual and contextual factors, with a special focus on the latency of rehabilitation start after hospital admission.

The study protocol complements measures of functioning with the indicators used in the registration form for clinical characterization cases disseminated by the World Health Organization: in doing so, the authors aim to support the global project of providing Member States with a standardized approach to collect clinical data.

Study objectives Primary Objective: To describe the emerging functional impairments in patients hospitalized for SARS-COV-2 infection (COVID-19), and monitor their course and impact on activities and participation up to 12 months of onset Secondary Objective: To search for predictive factors of recovery, among the pre-existing and emerging individual and context-related ones. Particular attention will be paid to the presence and latency of rehabilitation delivery after hospital admission, describing the functional evolution of subjects who received rehabilitation since the acute phase, compared to those who did not.

MATERIALS AND METHODS. Study Design. Prospective observational study with 12-month follow-up. Total study duration: 18 months Population. Adults, male and female, admitted to the University Hospital "Ospedali Riuniti of Ancona" (UH-ORA) from March 1st, 2020 for the management of acute COVID-19 infection, able to provide written or oral informed consent. The only exclusion criterion will be the lack of information concerning clinical data regarding the management in the acute ward.

Data collection: A paper CRF and an eCRF will be implemented to record patients' data

* Clinical, laboratory and instrumental data collected in the acute phase will be retrieved, retrospectively, from patients' clinical records.
* Data concerning function impairments, activity limitations and participation restrictions will be collected through direct assessment carried out by the rehabilitation team at the enrollment, on the first referral of the patient for counseling (T0) and at hospital discharge (Td) (for those who will receive rehabilitation in the acute ward), as well as at 3 , 6 and 12 months of COVID-19 diagnosis (T3, T6, T12). Patient reported outcomes will be assessed through questionnaires and interviews, also delivered by telephone or video-consultation.

The primary endpoint is the change in the overall health status observed at enrolment (T0), compared to the pre-COVID-19 condition, and its evolution at 3, 6 and 12 months. To this aim, we will assess:

* independence in activities of daily living (ADLs), by the modified Rankin scale. The modified Rankin scale is a rapid and validated measure of global independence in ADL with a score ranging from 0 (no disability) to 5 (bedridden). To assess changes, the pre-COVID mod. Rankin scale score, retrospectively ascertained, will be compared to the scores prospectively collected at enrolment and at 3, 6 and 12 months
* walking performance, by the Walking Handicap scale (WHS). The Walking Handicap scale is a quick and validated measure of walking performance, with a score ranging from 1 (Physiological walker: Walks for exercise only either at home or in parallel bars during physical therapy) to 6 (Community walker: Independent in all home and community activities. Can accept crowds and uneven terrain. Demonstrates complete independence in shopping centers). To assess changes, the pre-COVID WHS score, retrospectively ascertained, will be compared to the scores prospectively collected at 3, 6 and 12 months
* health-related quality of life perception, by the 36-Item Short Form Survey (SF-36). SF-36 is a widespread validated scale assessing patient-reported changes in health-related well-being perception over the last 4 weeks. SF-36 scores will be collected at 3, 6 and 12 months.

The secondary endpoint is the identification of the predictors of functional recovery at 3, 6 and 12 months, among the pre-existing and emerging individual and context-related factors.

The following explanatory variables will be considered:

* Pre-existing individual factors: age, gender, blood type, nutritional status, comorbidity (Modified Cumulative Illness Rating Scale - CIRS), life habits and pre-existing disability (modified Rankin Scale and Walking Handicap scale in pre-COVID phase)
* Emerging individual factors: severity of COVID-19 on admission to the acute ward, severity of pneumonia during hospitalization (according to Li et al 2020), blood chemistry (e.g. levels of interleukine, albumin, creatinine, CRP), pulmonary thromboembolism, neurologic complications, swallow disorders in the acute phase; severity of body function impairment and activity limitation on enrolment (as measured by the Trunk control test-TCT, Standing Balance-SB, Functional Ambulation Category-FAC, modified Barthel index- mBI, Montreal Cognitive Assessment-MoCA)
* Emerging context-related factors: drug treatment in the acute phase (e.g. ACE inhibitors, Angiotensin II receptor blockers, Nonsteroidal anti-inflammatories, Antivirals, heparin), procedures adopted in the ICU (prone positioning, tracheostomy, support for ventilation, ECMO, Renal replacement therapy or dialysis, Inotropes/vasopressors), rehabilitation delivery in the acute ward and latency from hospital admission to rehabilitation start.

Clinical-functional evaluations will be carried out at the following time-points:

T0 = on enrolment Td = discharge from the acute ward (only for subjects who are enrolled during their stay in the acute ward) T3, T6, T12 = three, six and 12 months after hospital admission due to COVID-19 infection.

After discharge from hospital, the assessments will be carried out in the outpatient laboratory; in case of mobility restrictions, questionnaires will be delivered and interviews will be conducted by telephone or by video consulting.

Sample size and data analysis. Given the nature of the study, a formal calculation of the sample size was not made. The enrolment of at least 100 subjects is estimated based on COVID-19 incidence in the catchment population of the UH-ORA.

A descriptive analysis will be conducted on the collected variables using point estimates and variability measures for quantitative variables or absolute and relative frequencies for category variables.

A multivariate model will be constructed to extrapolate predictors of poor recovery at 12 months (i.e. Delta T12-T0 on modified Rankin score : >1), by adjusting for potential confounders. After checking for the normal distribution of quantitative measures, the analysis of variance (ANOVA) for repeated measures will be applied to analyze the distribution of functional outcome measures, at 3, 6 and 12 months, among those who received rehabilitation in the acute phase, respect to those who did not.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years,
* any gender,
* COVID-19 diagnosis: positive oro-pharyngeal swab for SARS-COV-2
* admitted to the University Hospital "Ospedali Riuniti of Ancona" (UH-ORA) from March 1st, 2020 for the management of acute COVID-19,
* able to provide written or oral informed consent.

Exclusion Criteria:

* the lack of information concerning clinical data regarding the management in the acute ward.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults, male and female, admitted to the University Hospital "Ospedali Riuniti of Ancona" (UH-ORA) from March 1st, 2020 for the management of acute COVID-19 infection, able to provide written or oral informed consent. The only exclusion criterion will be the lack of information concerning clinical data regarding the management in the acute ward.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from pre-COVID-19 condition in ADL independence on the mod. Rankin scale score at the enrolment (T0) assessment, at 3, 6 and 12 months | Pre-COVID status, at enrolment and at 3, 6 12-month follow-up
  mod. Rankin scale is a rapid and validated measure of global independence in ADL with a score ranging from 0 (no disability) to 5 (bedridden).
  Change= pre-COVID mod. Rankin scale score (retrospective data) - mod. Rankin scale score prospectively collected at the enrolment (T0) and at 3, 6 and 12 months
Change from pre-COVID-19 condition in walking performance on the Walking Handicap scale (WHS) at 3, 6 and 12 months | Pre-COVID status , and 3, 6 12-month follow-up
  The Walking Handicap scale is a quick and validated measure of walking performance, with a score ranging from 1 (Physiological walker: Walks for exercise only either at home or in parallel bars during physical therapy) to 6 (Community walker: Independent in all home and community activities. Can accept crowds and uneven terrain. Demonstrates complete independence in shopping centers).
  Change= pre-COVID WHS (retrospective data) - WHS score prospectively collected at 3, 6 and 12 months
Patient-reported health-related well-being perception on the 36-Item Short Form Survey - SF-36 at 3, 6 12 months follow-up | 3, 6 and 12-month follow-up
  SF-36 is a widespread validated scale assessing patient-reported changes in health-related well-being perception over the last 4 weeks

SECONDARY OUTCOMES:
Change in global ADL disability on modified Barthel Index (mBI), from the enrolment (T0), at 3, 6 12 months follow-up | the enrolment (T0) assesssment and 3, 6 and 12-month follow-up
  The mBI is a validated measure of physical disability widely used to assess individual behavior in activities of daily living for patients with disabling conditions. It measures what patients do in practice. Score assignment can be made without any previous formal training.
  Change = mBI score at the enrolment (T0) assessment - mBI score at 3, 6 and 12-month follow-up
Change in walking capacity on Functional Ambulation Category (FAC), from the enrolment (T0) assessment, at 3, 6 12 months follow-up | Pre-COVID status, the enrollment (T0) assessment and 3, 6 12-month follow-up
  FAC is a validated measures of gait capacity with a score ranging from 0 (unable to walk) to 5 (able to walk independently in any environment)
  Change= pre-COVID FAC score (retrospective data) - FAC score prospectively collected at the enrolment (T0) assessment and at 3, 6 and 12 months
Change in cognitive abilities on the Montreal Cognitive Assessment (MoCA) from the enrollment (T0) assessment, at 3, 6 12 months follow-up | the enrollment (T0) assessment and 3, 6 and 12-month assessment follow-up
  The MoCA is a cognitive screening test designed to assist health professionals in the detection of mild cognitive impairment. It is especially sensitive at detecting dysfunctions in executive strategies.
  Change = MoCA score at the enrollment (T0) - MoCA score at 3, 6 and 12-month follow-up
Change in patient-reported pain on Numerical Rating Scale from the enrollment (T0) assessment, at 3, 6 12 months follow-up | the enrollment (T0) and 3, 6 and 12-month assessment follow-up
  Pain NRS is a widespread validate assessment tool measuring pain perception with a score ranging from 0 (no pain), to 10 (worst ever pain).
  Change= NRS score at the enrollment (T0) assessment - NRS score at 3, 6 and 12-month follow-up
Change in swallow abilities on Dysphagia Outcome Severity Scale (DOSS) from the first functional assessment in acute care, at 3, 6 12 months follow-up | the enrollment (T0) assessment and 3, 6 and 12-month assessment follow-up
  DOSS is a simple, easy-to-use, 7-point scale developed to systematically rate the functional severity of dysphagia based on objective assessment, with a score ranging from 1 (severe dysphagia: Non Per oral nutrition) to 7 ( Full per oral nutrition).
  Change= DOSS score at enrolment (T0) - DOSS score at 3, 6 and 12-month follow-up
Change in endurance on 6-Minutes Walking Test (6MWT) from the enrolment (T0) assessment, at 3, 6 12 months follow-up | the enrolment (T0) and 3, 6 and 12-month assessment follow-up
  6MWT is a validated and synthetic measure of endurance influenced by cardio-respiratory and motor function impairment.
  Change = 6MWT on enrolment (T0) - 6MWT score at 3, 6 and 12-month follow-up
Change in mood status on Beck Depression Inventory (BDI) from the enrolment (T0) assessment, at 3, 6 and 12 month follow-up | enrolment (T0) assessment and 3, 6 and 12-month assessment follow-up
  The BDI is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression.
  Change = BDI on enrolment (T0) assessment - BDI score at 3, 6 and 12-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Maria Gabriella Ceravolo, MD PhD, Study Director — Dep. of Experimental and Clinical Medicine - University Politecnica delle Marche
Locations (1):
- Neurorehabilitation Clinic, University Hospital Ospedali Riuniti di Ancona, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No
The research results will be made available through indexed Journals as scientific publication.

REFERENCES:
- [Background] Ceravolo MG, de Sire A, Andrenelli E, Negrini F, Negrini S. Systematic rapid "living" review on rehabilitation needs due to COVID-19: update to March 31st, 2020. Eur J Phys Rehabil Med. 2020 Jun;56(3):347-353. doi: 10.23736/S1973-9087.20.06329-7. Epub 2020 Apr 22. PMID 32316718
- [Background] Andrenelli E, Negrini F, de Sire A, Arienti C, Patrini M, Negrini S, Ceravolo MG; International Multiprofessional Steering Committee of Cochrane Rehabilitation REH-COVER action. Systematic rapid living review on rehabilitation needs due to COVID-19: update to May 31st, 2020. Eur J Phys Rehabil Med. 2020 Aug;56(4):508-514. doi: 10.23736/S1973-9087.20.06435-7. Epub 2020 Jun 16. PMID 32539312
- [Background] de Sire A, Andrenelli E, Negrini F, Negrini S, Ceravolo MG. Systematic rapid living review on rehabilitation needs due to COVID-19: update as of April 30th, 2020. Eur J Phys Rehabil Med. 2020 Jun;56(3):354-360. doi: 10.23736/S1973-9087.20.06378-9. Epub 2020 May 15. PMID 32408729
- [Background] Ahmad I, Rathore FA. Neurological manifestations and complications of COVID-19: A literature review. J Clin Neurosci. 2020 Jul;77:8-12. doi: 10.1016/j.jocn.2020.05.017. Epub 2020 May 6. PMID 32409215
- [Background] Yang LL, Yang T. Pulmonary rehabilitation for patients with coronavirus disease 2019 (COVID-19). Chronic Dis Transl Med. 2020 May 14;6(2):79-86. doi: 10.1016/j.cdtm.2020.05.002. eCollection 2020 Jun. PMID 32411496
- [Background] Brugliera L, Spina A, Castellazzi P, Cimino P, Arcuri P, Negro A, Houdayer E, Alemanno F, Giordani A, Mortini P, Iannaccone S. Nutritional management of COVID-19 patients in a rehabilitation unit. Eur J Clin Nutr. 2020 Jun;74(6):860-863. doi: 10.1038/s41430-020-0664-x. Epub 2020 May 20. No abstract available. PMID 32433599
- [Background] Negrini S, Grabljevec K, Boldrini P, Kiekens C, Moslavac S, Zampolini M, Christodoulou N. Up to 2.2 million people experiencing disability suffer collateral damage each day of COVID-19 lockdown in Europe. Eur J Phys Rehabil Med. 2020 Jun;56(3):361-365. doi: 10.23736/S1973-9087.20.06361-3. Epub 2020 May 8. PMID 32383576
- [Background] Bartolo M, Intiso D, Lentino C, Sandrini G, Paolucci S, Zampolini M; Board of the Italian Society of Neurological Rehabilitation (SIRN). Urgent Measures for the Containment of the Coronavirus (Covid-19) Epidemic in the Neurorehabilitation/Rehabilitation Departments in the Phase of Maximum Expansion of the Epidemic. Front Neurol. 2020 Apr 30;11:423. doi: 10.3389/fneur.2020.00423. eCollection 2020. PMID 32425880
- [Background] Lew HL, Oh-Park M, Cifu DX. The War on COVID-19 Pandemic: Role of Rehabilitation Professionals and Hospitals. Am J Phys Med Rehabil. 2020 Jul;99(7):571-572. doi: 10.1097/PHM.0000000000001460. PMID 32371624
- [Background] Li H, Xue Q, Xu X. Involvement of the Nervous System in SARS-CoV-2 Infection. Neurotox Res. 2020 Jun;38(1):1-7. doi: 10.1007/s12640-020-00219-8. Epub 2020 May 13. PMID 32399719
- [Background] Valenzuela PL, Joyner M, Lucia A. Early mobilization in hospitalized patients with COVID-19. Ann Phys Rehabil Med. 2020 Jul;63(4):384-385. doi: 10.1016/j.rehab.2020.04.005. Epub 2020 May 18. No abstract available. PMID 32418848
- [Background] Stein J, Visco CJ, Barbuto S. Rehabilitation Medicine Response to the COVID-19 Pandemic. Am J Phys Med Rehabil. 2020 Jul;99(7):573-579. doi: 10.1097/PHM.0000000000001470. PMID 32433243
- [Background] Wang X, Xu H, Jiang H, Wang L, Lu C, Wei X, Liu J, Xu S. Clinical features and outcomes of discharged coronavirus disease 2019 patients: a prospective cohort study. QJM. 2020 Sep 1;113(9):657-665. doi: 10.1093/qjmed/hcaa178. PMID 32442308